CLINICAL TRIAL: NCT03312595
Title: Clinical Outcomes After Treatment With RestrataTM Wound Matrix in Diabetic Foot Ulcers (DFU) A Case Series of Initial Effectiveness and Safety Measures
Brief Title: Clinical Outcomes After Treatment With RestrataTM Wound Matrix in Diabetic Foot Ulcers (DFU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acera Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-RES-001
Record Dates: First submitted 2017-10-01; First posted 2017-10-18 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Restrata TM Wound Matrix (Other): Prospective, single armed, non-randomized study with direct assignment
  Interventions: Device: Restrata TM Wound Matrix

INTERVENTIONS:
Device: Restrata TM Wound Matrix — The RestrataTM Wound Matrix is a sterile, single use device intended for use in local management of wounds

SUMMARY:
The primary objective of this study is to determine the outcomes of patients who receive a certain type of skin substitute called RestrataTM Wound Matrix (Restrata™). Results of this study may be used to make decisions on whether to conduct additional studies on this particular wound matrix product. RestrataTM has been cleared by the Food and Drug Administration for use in certain types of ulcer treatments, including the type that will be part of this study (diabetic foot ulcers).

DETAILED DESCRIPTION:
Control Group: None (Utilize historical / published data on outcomes using standard of care)

Test Group: Treatment of DFUs with RestrataTM Wound Matrix

Study Type: Interventional

Study Design: Allocation: Non-randomized Endpoint Classification: Efficacy Intervention Model: Direct assignment Masking: Single Blind (Subject) Primary Purpose: Treatment

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 or older
* Patient's ulcer must be diabetic in origin, located at least in part on the plantar surface and larger than 1cm2 after the run-in period. Debridement will be done prior to randomization. Subject's informed consent for participating in this study, must be obtained prior to proceeding with sharp debridement
* Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
* Ulcer must be present for a minimum of four weeks before enrollment/randomization, with documented failure of prior treatment to heal the wound. A two-week run in period will precede enrollment/randomization in the trial to document the indolent nature of the patients selected
* Patient does not exhibit clinical signs / symptoms of infection upon gross observation (at least 3 of the following: pain, redness, purulence, exudate, temperature) or have been diagnosed with an active infection at time of screening
* Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study
* Patient has adequate control of diabetes, as demonstrated by one of the following within 30 days of screening:

  * HbA1c < 12%
  * Serum Creatinine < 3.0mg/dl
* Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days of the first screening visit:

  * Dorsum transcutaneous oxygen test (TcPO2) with results

    ≥30mmHg, OR
  * ABIs with results of ≥0.7 and ≤1.5, OR
  * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg

Exclusion Criteria:

* Patients presenting with an ulcer probing to bone (UT Grade IIIA-D)
* Patients whose index diabetic foot ulcers are greater than 25cm2
* Patient has an additional wound within 3cm of the study wound
* Patients not in reasonable metabolic control
* Patients with a known history of poor compliance with medical treatments
* Patients who have been previously enrolled into this study, or are presently participating in a clinical trial with DFU indications
* Patients with known or suspected local skin malignancy to the index diabetic ulcer
* Patients diagnosed with autoimmune connective tissues diseases
* Patients that have received a graft material on the study ulcer within the previous 30 days
* Patients who are pregnant or breast feeding
* Patients who are taking medications that are considered immune system modulator
* Study wound has closed > 30% over the two-week run-in period
* Patients with a known allergy to resorbable suture materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Associated Foot & Ankle Specialists, Phoenix, Arizona
  - Arizona Reginal Medical Research, Tucson, Arizona
  - SAVAHCS, Tucson, Arizona
  - Advanced Foot Care And Clinical Research Center, Fresno, California
  - Richard C. Galperin, DPM, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Restrata Wound Matrix: Prospective, single armed, non-randomized study with direct assignment
  Restrata Wound Matrix: The Restrata Wound Matrix is a sterile, single use device intended for use in local management of wounds
Period: Overall Study
Arm/Group | Restrata Wound Matrix
Started | 30
Completed | 24
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Restrata Wound Matrix
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — Population: Data not consistently reported for all patients
  Participants
    number analyzed (Participants) | 20
    <=18 years | 0
    Between 18 and 65 years | 19
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not consistently reported for all patients
  Participants
    number analyzed (Participants) | 20
    Female | 2
    Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Wound Closed
Description: from baseline at week 0 to 14 weeks
Time Frame: Up to 14 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Restrata Wound Matrix
Number analyzed (Participants) | 24
percentage of participants | 75

2. Secondary Outcome: Change in Wound Area From Baseline
Description: Wound area measurements will be made via tracing acetate every week for 14 weeks.
Time Frame: Baseline and weekly for up to 14 weeks
Measure: Mean (Standard Deviation); unit: % wound area change
Arm/Group | Restrata Wound Matrix
Number analyzed (Participants) | 24
% wound area change | 96 (10)

3. Secondary Outcome: Time to Wound Closure
Description: The number of weeks until complete closure is first identified will be determined for each patient who has been deemed completely closed within the 14 week treatment period.
Time Frame: Baseline up to 14 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Restrata Wound Matrix
Number analyzed (Participants) | 18
weeks | 6.4 (2.5)

ADVERSE EVENTS:
Time Frame: 3.5 months
Arm/Group | Restrata Wound Matrix
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 12/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restrata Wound Matrix (N=24)
Fever (General disorders) | 1 — Deemed not due to Restrata Wound Matrix.
Infection (General disorders) | 3 — Deemed not due to Restrata Wound Matrix.
Trauma (General disorders) | 2 — Deemed not due to Restrata Wound Matrix.
Osteomyelitis (General disorders) | 2 — Deemed not due to Restrata Wound Matrix.
Peripheral vascular disease (General disorders) | 1 — Deemed not due to Restrata Wound Matrix.
Blister (General disorders) | 2 — Deemed not due to Restrata Wound Matrix.
New ulcer (General disorders) | 1 — Deemed not due to Restrata Wound Matrix.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT03312595/Prot_SAP_001.pdf